CLINICAL TRIAL: NCT00188487
Title: MR Perfusion Imaging in Asthmatic Patients
Brief Title: Magnetic Resonance (MR) in Asthmatic Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no funding
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-0174
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Magnetic Resonance Imaging

INTERVENTIONS:
Device: magnetic resonance imaging (MRI) of the thorax

SUMMARY:
Asthma is a disease of small airways. Affected areas have reduced lung ventilation causing reflex vasoconstriction. MR perfusion imaging of the lungs is a sensitive method of imaging zonal lung perfusion.

DETAILED DESCRIPTION:
A cohort of 70 Asthmatic Patients and 10 controls, both sets of subjects have HRCT, MRI/A of the Thorax, and Pulmonary Function Tests to correlate the degree of pulmonary dysfunction with findings on imaging tests.

ELIGIBILITY:
Inclusion Criteria:

* All asthmatic patients are eligible.

Exclusion Criteria:

* Patients in whom MRI is contraindicated

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2005-09; Study Completion 2005-12

PRIMARY OUTCOMES:
The correlation of MR lung perfusion analysis with computed tomography (CT) findings and pulmonary function tests

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FRCP C, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada